CLINICAL TRIAL: NCT01896050
Title: A Prospective Assessment of Loss of Grip Strength by Baseline BMI in Breast Cancer Patients Receiving Adjuvant Third-generation Aromatase Inhibitors and Tamoxifen
Brief Title: Loss of Grip Strength, BMI, and Adjuvant Endocrine Therapy Breast Cancer
Acronym: LOGRIBMET
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Principal Investigator, Lynn Henry, Principal Investigator, University of Michigan Rogel Cancer Center
Other Study IDs: UMCC 2009.029
Record Dates: First submitted 2013-07-05; First posted 2013-07-11 (Estimated); Results first posted 2016-05-12 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer; Arthralgia; Obesity
Keywords: Joint pain; Grip strength; Hormone receptor positive breast cancer
MeSH Terms: conditions — Breast Neoplasms; Arthralgia; Obesity | interventions — Anastrozole; Letrozole; exemestane; Tamoxifen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood is being collected at baseline for DNA extraction. Serum is being collected at baseline and after 3, 6, and 12 months.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AI therapy: Subjects who started treatment with any of the three aromatase inhibitor (AI) medications
  Interventions: Drug: anastrozole, letrozole, exemestane
- Tamoxifen: Subjects who started treatment with tamoxifen
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: anastrozole, letrozole, exemestane — Patients were treated with one of the listed anti-hormonal medications for up to one year
  Other Names: Arimidex, Femara, Aromasin
  Groups: AI therapy
Drug: Tamoxifen — Patients were treated with tamoxifen for up to one year
  Other Names: Novaldex
  Groups: Tamoxifen

SUMMARY:
Early stage hormone receptor positive breast cancer is typically treated with adjuvant endocrine therapy in order to decrease risk of breast cancer recurrence and to improve overall survival from the disease. Typical agents used for treatment include tamoxifen and the aromatase inhibitors. In postmenopausal women, aromatase inhibitor therapy is increasingly common because it is associated with fewer long-term serious toxicities compared to tamoxifen. However, aromatase inhibitors cause arthralgias in 40-50% of patients, which can influence adherence to therapy and can lead to treatment discontinuation in a minority of cases. The mechanism underlying development of this toxicity remains unclear, and predictors of who will develop these symptoms remain undefined. Initial reports suggest that grip strength decreases during aromatase inhibitor therapy, and that body-mass index may influence development of this symptom. Therefore, this longitudinal study has been developed to determine change in grip strength over time in women treated with aromatase inhibitors and tamoxifen, as well as to identify potential associations between change in grip strength and BMI. Patient self-reported symptoms will also be collected. A total of 115 women with early stage breast cancer who are initiating therapy with either an aromatase inhibitor or tamoxifen will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Stage 0-III breast cancer who are scheduled to receive endocrine therapy with tamoxifen or an aromatase inhibitor
* All prior surgery and chemotherapy should be complete
* Age 18 and above and postmenopausal

Exclusion Criteria:

* Major rheumatologic disorders
* Concomitant sex hormone containing drugs or Leutinizing Hormone Releasing Hormone agonist therapy
* For those subjects initiating treatment with an aromatase inhibitor, prior tamoxifen within 4 weeks of enrollment
* For those subjects initiating treatment with tamoxifen, prior aromatase inhibitor within 4 weeks of enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with hormone receptor positive breast cancer who are initiating therapy with either an aromatase inhibitor or tamoxifen.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2009-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Henry, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AI Therapy | Tamoxifen
Started | 93 | 22
Completed | 55 (This includes only patients who remained on the same aromatase inhibitor medication for 12 months) | 20
Not Completed | 38 | 2
Not completed — Adverse Event | 37 | 2
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AI Therapy | Tamoxifen | Total
Number analyzed (Participants) | 93 | 22 | 115
Age, Continuous [Median (Full Range); unit: years] | 62 [41 to 79] | 61.5 [44 to 69] | 62 [41 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 22 | 115
  Male | 0 | 0 | 0
Body-mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.4 (7.1) | 29 (7) | 30.1 (7.1)
Waist-hip ratio [Mean (Standard Deviation); unit: ratio] | 0.91 (0.09) | 0.92 (0.12) | 0.91 (0.09)
Maximum grip strength, right hand [Mean (Standard Deviation); unit: kPa] | 57.5 (11.7) | 56.4 (10.9) | 57.3 (11.5)
Maximum grip strength, left hand [Mean (Standard Deviation); unit: kPa] | 54.8 (10.9) | 53.7 (10.7) | 54.6 (10.8)
Average pain [Mean (Standard Deviation); unit: units on a scale] — Patients reported pain on a 0-10 visual analog scale, with 0 being no pain and 10 being worst pain imaginable.
  units on a scale | 2.3 (2.1) | 2.4 (1.9) | 2.3 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Change in Body Mass Index on Change in Grip Strength With Aromatase Inhibitor Therapy
Description: Change in BMI between baseline and 12 months of endocrine therapy
Time Frame: baseline and 12 months
Population: These data only include patients who completed a full 12 months of treatment with either an aromatase inhibitor or tamoxifen and had grip strength data at both baseline and 12 months. Patients could have switched from one aromatase inhibitor to another. Those patients who discontinued treatment prior to the 12 month period were excluded.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | AI Therapy | Tamoxifen
Number analyzed (Participants) | 71 | 18
kg/m^2 | -0.15 (5.70) | 2.44 (6.11)
Statistical Analysis 1: Comparison: AI Therapy vs Tamoxifen; Compare difference in change in body mass index between baseline and 12 months between aromatase inhibitor- and tamoxifen-treated patients; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: AI Therapy; Examine association between change in body mass index and change in grip strength with aromatase inhibitor therapy. For the primary outcome, linear regression was used for analysis with change of grip strength as response variable. In the original statistical analysis plan only aromatase inhibitor-treated patients were to be included in this analysis. This analysis was not performed on the tamoxifen group because it isn't clinically relevant; Test type: Superiority or Other; p = 0.4262, Regression, Linear; BMI squared = -0.01845, Standard Error of Mean 0.02308

2. Secondary Outcome: Effect of Medication on Change in Grip Strength
Description: Effect of either aromatase inhibitor or tamoxifen therapy on change in grip strength between baseline and 12 months
Time Frame: baseline and 12 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | AI Therapy | Tamoxifen
Number analyzed (Participants) | 93 | 22
percent change | -7.0 (15.9) | 0.6 (10.2)
Statistical Analysis 1: Comparison: AI Therapy vs Tamoxifen; Comparison of change in maximum grip strength between baseline and 12 months for aromatase inhibitor-treated versus tamoxifen-treated patients; Test type: Superiority or Other; p = 0.032, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Association Between Baseline Body Mass Index and Discontinuation of Aromatase Inhibitor Therapy Within the First 12 Months
Description: Associations between baseline BMI and whether or not aromatase inhibitor-treated patients discontinued treatment by 12 months. In the original statistical analysis plan, it was only intended to examine the association with aromatase inhibitor-treated patients, and not tamoxifen-treated patients. The numbers below reflect the number of patients in each group who discontinued initial endocrine therapy within the first 12 months of treatment
Time Frame: baseline and 12 months
Measure: Number; unit: participants
Groups:
- Aromatase Inhibitor: Aromatase inhibitor-treated patients
- Tamoxifen: Tamoxifen-treated patients
Arm/Group | Aromatase Inhibitor | Tamoxifen
Number analyzed (Participants) | 93 | 22
participants | 37 | 2
Statistical Analysis 1: Comparison: Aromatase Inhibitor; Association between baseline body mass index and discontinuation of aromatase inhibitor therapy. The original statistical analysis plan only called for analyzing the aromatase inhibitor-treated patients, not the tamoxifen-treated patients; Test type: Superiority or Other; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.92 to 1.04]

ADVERSE EVENTS:
Time Frame: 12 months
Description: only unexpected serious adverse events were collected
Arm/Group | AI Therapy | Tamoxifen
Serious Adverse Events (participants affected / at risk) | 1/93 | 0/22
Other Adverse Events (participants affected / at risk) | 37/93 | 2/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AI Therapy (N=93) | Tamoxifen (N=22)
death (General disorders) | 1 (1) | 0 (0) — one patient died during study participation of reasons unrelated to study participation or AI therapy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AI Therapy (N=93) | Tamoxifen (N=22)
symptom leading to treatment discontinuation (General disorders) | 37 (37) | 2 (2) — For expected toxicities, we only collected information about whether a patient felt her symptoms were bothersome enough to stop treatment, not treatment about the individual symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No